CLINICAL TRIAL: NCT01772394
Title: Cognitive Remediation Therapy Effectiveness in Anorexia Nervosa: a Multicenter Randomized Clinical Study
Brief Title: Cognitive Remediation Therapy in Anorexia Nervosa
Acronym: TreCogAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCB-2011-A01280-41; P091123 (Other: AP-HP)
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Teenager; Young Adult; Hospitalized; Anorexia Nervosa (DSM-IV Revised Criteria)
Keywords: Anorexia Nervosa; Cognitive remediation therapy; Randomized clinical trial
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Remediation Therapy (CRT) (Active Comparator): Active : CRT
  Interventions: Behavioral: Cognitive Remediation Therapy
- Sham Therapy (ST) (Sham Comparator): Sham : ST
  Interventions: Behavioral: Sham Therapy

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy — Cognitive remediation therapy (CRT) is an intensive training cognitive therapy that encourages people to reflect on and try to modify the way they think, with a particular focus on improving cognitive flexibility. It is a manualised therapist-led intervention consisting of multiple versions of a variety of tasks and mental exercises that address the difficulties in flexibility and holistic processing. CRT is an individual 10-sessions long program (2 sessions per week).
  Other Names: CRT
  Arms: Cognitive Remediation Therapy (CRT)
Behavioral: Sham Therapy — The Sham therapy (ST) has been designed to match the CRT format: an individual manualised therapist-led 10-sessions long program (2 sessions per week). ST sessions have been designed so as to avoid set-shifting and central coherence training. Rather, ST is a manualised sham intervention consisting of multiple exercises on 3 domains: soft physical activity, emotional expression recognition and interpersonal functioning.
  Other Names: ST
  Arms: Sham Therapy (ST)

SUMMARY:
"Clinicians from the Maudsley (IoP, London, UK) have specifically tailored a cognitive remediation therapy (CRT) for treating Anorexia Nervosa (AN). It is an intensive manualised training cognitive therapy which addresses the difficulties in flexibility and holistic processing that have been incriminated in AN. CRT has been found to improve AN's neuropsychological functioning and short term outcome. To our knowledge, no French speaking country has tested its effectiveness. Moreover, the question whether it is efficient for both anorexic restrictive and anorexic binge-purging patients remains unanswered.

The aim of the present study is to determine if CRT in AN adolescents and young adults has a favourable impact on cognitive functioning and clinical status. We will also explore whether the impact of CRT is similar in both anorexic restrictive and binge-purging subtypes. There will also be an Historical Control Group of patients, sixty, who received traditional medical interventions in a specialized inpatient unit for eating disorders (i.e., EVHAN study)."

DETAILED DESCRIPTION:
"Several studies have documented that patients with Anorexia Nervosa (AN) display a trait of cognitive inflexibility (e;g., poor set-shifting performances on the Trail Making Task B), i.e. an inability to move flexibly back and forth between tasks, operations, or mental sets which allows for the adaptation of behaviour in response to changing demands within the environment. This cognitive inflexibility can be observed both during the acute phase of the illness and after weight restoration, and has been found to predict negative treatment outcomes. 'Weak central coherence' is another skill which is particularly problematic in AN. It refers to a cognitive style in which information remains fragmented as opposed to integrated, with processing occurring at the level of 'detail' as opposed to 'whole'. AN patients exhibit this detail focussed information-processing style (e.g., as measured by the Embedded Figures Test). To treat these difficulties, clinicians from the Institute of Psychiatry (London, UK) have specifically tailored a treatment for AN. Cognitive remediation therapy (CRT) is an intensive training cognitive therapy that encourages people to reflect on and try to modify the way they think, with a particular focus on improving cognitive flexibility. It is a manualised therapist-led intervention consisting of multiple versions of a variety of tasks and mental exercises that address the difficulties in flexibility and holistic processing. CRT is a 10-sessions long program that has been found to improve AN's neuropsychological functioning and short term outcome. To our knowledge, no French speaking country has tested its effectiveness. Moreover, the question whether it is efficient for both anorexic restrictive and anorexic binge-purging patients remains unanswered.

To address these issues, we designed a multicenter randomized clinical trial on the effectiveness of CRT in AN adolescents and young adults.

Main hypothesis: AN patients treated with CRT present a better clinical status than those treated by a control therapy.

Recruitment and Procedure: 120 female adolescents or young adults [15-40 years old] AN (60 Anorexic Restrictive; 60 Anorexic Binge-Purging) will be recruited among the patients of specialized ED care units of three hospitals: PAUL BROUSSE, INSTITUT MUTUALISTE MONTSOURIS, COCHIN-MAISON DE SOLENN. In each group of AN subtype, the patients will be randomly allocated to one of the two treatment arms: CRT or Sham Therapy (ST). Each therapy is manualised and includes 10 sessions over a period of 5 weeks (2 sessions/week). All the patients will be assessed just prior the beginning and after the end of the CRT/ST, at 6 months and 1 year of follow-up."

ELIGIBILITY:
Inclusion Criteria:

* female;
* 15-40 years old;
* hospitalised for a diagnosis of Anorexia Nervosa (DSM-IV Revised criteria) in one of the three departments participating in this research ;
* fluent in French;
* who provide their informed consent (or as far as possible their parents for those under 18).

Exclusion Criteria:

* previous history of neurological disorders;
* actual substance use disorder;
* schizophrenia;
* presenting a related somatic illness (diabetes, Crohn's disease, metabolic illness) or a life-threatening condition.

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Neuropsychological functioning:Wisconsin Sorting Card Test (WSCT) | 1 week post-therapy
  The WSCT are two neuropsychological tests that have been consistently used to highlight poor set-shifting skills in Anorexia nervosa.
Clinical status Evaluation:Morgan and Russell Global Outcome Assessment Scale (GOAS); | up to 1 year of follow-up
  The Global Outcome Assessment Schedule (GOAS; Morgan & Hayward, 1998) is a standard measure of outcome in eating disorders; it includes 14 subscales evaluating five dimensions: (A) Food Intake and body weight ; (B) Menstrual status; (C) Mental state ; (D) Psychosexual state ; (E) Socioeconomic status and social functioning.

SECONDARY OUTCOMES:
Central coherence | 1 week post-therapy
  Central coherence: Rey figure;
Nutritional status | 1 week post-therapy
  body mass index
Nutritional status | 6 months of follow-up
  body mass index
Nutritional status | 1 year of follow-up
  body mass index
Self-reported eating disorders symptoms | 1 week post-therapy
  Eating Disorder Examination Questionnaire and Body Shape Questionnaire
Self-reported eating disorders symptoms | 1 year of follow-up
  Eating Disorder Examination Questionnaire and Body Shape Questionnaire
Self-reported Cognitive style; | 1 week post-therapy
  Detail and Flexibility Questionnaire
Self-reported Cognitive style; | 1 year of follow-up
  Detail and Flexibility Questionnaire
Self-reported treatment satisfaction | 1 week post-therapy
  Helping Alliance Questionnaire and Patient Satisfaction Questionnaire
Self-reported motivation to change | 1 week post-therapy
  the Maudsley motivation to change questionnaire
Self-reported motivation to change | 6 months of follow-up
  the Maudsley motivation to change questionnaire
Self-reported motivation to change | 1 year of follow-up
  the Maudsley motivation to change questionnaire
Self-reported self-esteem | 1 week post-therapy
  Rosenberg self-esteem Questionnaire
Self-reported self-esteem | 1 year of follow-up
  Rosenberg self-esteem Questionnaire
Flexibility evolution : Trail Making Test (TMT) | 1 week post-therapy
  Neuropsychological functioning

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie BERTHOZ, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Damien RINGUENET, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Clinique Villa Montsouris, Paris
  - Institut Mutualiste Monsouris, Paris
  - Maison de Solenn, Paris
  - Assistance Publique - Hôpitaux de Paris, Hôpital Paul Brousse, Villejuif

REFERENCES:
- [Derived] Maria AS, Barry C, Ringuenet D, Falissard B, Group T, Berthoz S. Subjective cognitive rigidity and attention to detail: A cross-cultural validation of the Detail and Flexibility Questionnaire (DFlex) in a French clinical sample. J Clin Exp Neuropsychol. 2020 Dec;42(10):1059-1071. doi: 10.1080/13803395.2020.1842333. Epub 2020 Dec 4. PMID 33274668
- [Derived] Maria AS, Bourdier L, Duclos J, Ringuenet D, Berthoz S. Psychometric properties of the French version of a scale measuring perceived emotional intelligence : the Trait Meta-Mood Scale (TMMS). Can J Psychiatry. 2016 Oct;61(10):652-62. doi: 10.1177/0706743716639936. Epub 2016 Mar 28. PMID 27310229